CLINICAL TRIAL: NCT00399334
Title: Study PROFILe3: Clinic Observations Profile of Relapse and Readmission in Emergency/Acute Settings: Epidemiologic Survey in Schizophrenic Patients
Brief Title: PROFILe3: Epidemiologic Survey in Patients With Schizophrenia or Schizoaffective Disorders
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR010609
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Schizoaffective; relapse; risk factors; Observational study; Antipsychotic medication
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: antipsychotic medications

INTERVENTIONS:
Drug: antipsychotic medications — as prescribed

SUMMARY:
The purpose of this study is to evaluate epidemiological characteristics of patients that experience relapse and need an admission in psychiatric acute units across Spain.

DETAILED DESCRIPTION:
Long-term treatment in schizophrenia begins in acute hospitalization. However inadequate treatment options in non-compliant patients discharged from acute inpatient settings are often leading to recidivism and frequent re-hospitalization. The objective of this epidemiologic survey is to evaluate epidemiological characteristics of relapse and readmission in acute psychiatric units. If long-term treatment in schizophrenia begins in acute hospitalization the use of the new long-acting injectable antipsychotics after an acute psychotic episode as a standard maintenance medication could prevent relapse and readmissions. This is a pharmaco-epidemiological study, which collects structured safety data and it is carried out in Spain. All data collected will be cross-sectional or retrospective and will include the following: demographic data, diagnosis, psychiatric history and co-morbidities, hospitalization record (previous 3 years), treatment record and physician's opinion on patient's treatment compliance. The primary objectives are to evaluate epidemiological characteristics of patients that experience relapse and need an admission in psychiatric acute units across Spain, to determine the most important risk factors which predicts the number of hospital re-admissions and to identify the impact of the clinical profile of patients with schizophrenia, and schizoaffective/schizophreniform disorders who suffer relapses. The second objective is to describe the clinical decisions made by psychiatrist regarding therapeutic approach according to the previous characteristics of the patient. as prescribed

ELIGIBILITY:
Inclusion Criteria:

* Patients with Schizophrenia or Schizoaffective disorder with a diagnosis over 2 years and that are hospitalized in a Short-Term Psychiatric Hospitalization Unit or Acute Unit

Exclusion Criteria:

* Patients with psychiatry pathology other than Schizophrenia or schizoaffective disorder
* Patients with Schizophrenia or Schizoaffective disorder with a diagnosis less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Schizophrenia or Schizoaffective disorder with a diagnosis over 2 years that are hospitalized in a Short-Term Psychiatric Hospitalization Unit or Acute Unit.
Sampling Method: Non-Probability Sample
Enrollment: 1607 (Actual)
Dates: Start 2005-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Determine the epidemiological characteristics of patients that experience relapse and need an admission in psychiatric acute units across Spain | All data is collected in just one visit (i.e. cross-sectional and retrospective data)

SECONDARY OUTCOMES:
Describe the clinical decisions made by psychiatrist regarding therapeutic approach according to the previous characteristics of the patient. | 1 visit (cross-sectional study)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Epidemiological study to analyze the clinical profile of patients with schizophrenia in short-stay psychiatric hospitalization units — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=285&filename=CR010609_CSR.pdf